CLINICAL TRIAL: NCT05222048
Title: Endoscopy Needs of People in Suichang County
Brief Title: Endoscopy Needs of People in Suichang County, Lishui City, Zhejiang Province, China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: Suichang-2021(38)
Record Dates: First submitted 2021-12-29; First posted 2022-02-03 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2021-12

CONDITIONS: Gastrointestinal Endoscopy
Keywords: Gastrointestinal endoscopy, demand analysis,

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
With the improvement of people's health awareness, more and more people realize the importance of endoscopy. Compared with other imaging methods (such as gastrointestinal contrast, abdominal ultrasound, CT, MR, nuclear medicine, etc.), in addition to the diagnosis of diseases, endoscopy also has obvious advantages in obtaining specimens for further pathological examination. However, the pain and discomfort caused by endoscopy have discouraged many people and even missed the opportunity for early diagnosis. At present, painless endoscopy can improve this kind of situation, but everyone has various doubts about it. In order to accurately understand and grasp the needs of people in Suichang County for gastrointestinal endoscopy, so as to better carry out gastrointestinal endoscopy/screening/diagnosis and treatment work in the future, we designed this demand survey.

ELIGIBILITY:
Inclusion Criteria:

* All people who come to the endoscopy center for gastrointestinal endoscopy, as well as those who may have gastrointestinal endoscopy in outpatient clinics, ward patients and other social groups, and are willing to participate in the questionnaire survey.

Exclusion Criteria:

* People who cannot cooperate, are unconscious, or who are unwilling to participate in questionnaire surveys.

Max Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Permanent resident population above 14 years old in Suichang County, excluding foreign nationals.
Sampling Method: Probability Sample
Enrollment: 1061 (Estimated)
Dates: Start 2021-10-12 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Individual choice of anesthesia during gastrointestinal endoscopy | 1 day
  We will use the questionnaire to assess this outcome measure.
  Part of the questionnaire is as follows:
  1. What type of endoscopy was done this time (or last time)? [indefinite multiple choice]
     * Ordinary gastroscopy
     * Ordinary colonoscopy
     * Painless gastroscopy
     * Painless colonoscopy
     * Painless gastroenteroscopy
  2. Which type will you choose for your next gastroenteroscopy? [Multiple choice]
     * Painless
     * A single gastroscope is normal, and a single colonoscope is painless
     * A single gastroscope is painless, and a single colonoscope is normal
     * Under no circumstances anesthesia
     * Normal, but if performed together with gastroenteroscopy, it is still painless

SECONDARY OUTCOMES:
Individual attitude towards gastrointestinal endoscopy follow-up | 1 day
  We will also use the questionnaire to assess this outcome measure.
  Part of the questionnaire is as follows:
  Will you have a gastroenteroscopy next time? [single choice]
  * I will be reviewed regularly.
  * I will do it when I have symptoms.
  * It is really necessary to reconsider doing it.
  * I never want to do it again.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastroenterology, Suichang People's Hospital, Lishui, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided